CLINICAL TRIAL: NCT01494636
Title: A Two Part Study to Investigate the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2339345 in Healthy Subjects. Part A: an Open Label, Dose Escalating, Rinse, Gargle and Spit Study. Part B: a Randomised, Double-blind, Placebo Controlled, Inhaled Dose Escalating Study Using Nebulised Lidocaine for Blinding Purposes.
Brief Title: The Safety, Tolerability, PK and PD of GSK2339345 in Healthy Subjects
Acronym: FTIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115419
Record Dates: First submitted 2011-11-17; First posted 2011-12-19 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Cough
Keywords: Capsaicin Challenge; Pharmacodynamics; Safety; Pharmacokinetics; Oral GSK2339345; Tolerability; FTIH; Chronic Cough
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Solutions; Sodium Chloride; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK2339345 (solution) (part A) (Experimental): Part A
  Interventions: Drug: GSK2339345 (solution)
- GSK2339345/ Placebo/ Lidocaine (nebulised) (part B) (Experimental): Part B
  Interventions: Drug: GSK2339345 (nebulised); Drug: Placebo (0.9% sodium chloride solution); Drug: Lidocaine

INTERVENTIONS:
Drug: GSK2339345 (solution) — 3, 6, 15, 30, 60 and 120 micrograms (proposed doses). 2 alternating cohorts of 6 subjects. Each subject to receive 3 ascending doses with washout of at least 48 hours between doses. Rinse, Gargle and Spit.
  Arms: GSK2339345 (solution) (part A)
Drug: GSK2339345 (nebulised) — 25, 100, 250, 1000 and 2000 micrograms (proposed doses). Subjects randomised to receive three ascending doses (with each dose given on two consecutive days). Washout of at least 6 days between treatment periods. Nebulised.
  Arms: GSK2339345/ Placebo/ Lidocaine (nebulised) (part B)
Drug: Placebo (0.9% sodium chloride solution) — Administered on Day 1 of one of the treatment periods in part B. Randomised. Nebulised.
  Arms: GSK2339345/ Placebo/ Lidocaine (nebulised) (part B)
Drug: Lidocaine — 40mg dose. Administered on Day 2 of one of the treatment periods in part B. Randomised. Nebulised.
  Arms: GSK2339345/ Placebo/ Lidocaine (nebulised) (part B)

SUMMARY:
This is a First Time in Human (FTIH) study for the sodium channel inhibitor, GSK2339345. The study is split into two parts. Part A will assess the safety and tolerability of the new drug. Part B will assess safety and tolerability as well as the effect of GSK2339345 on induced cough.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) effects of GSK2339345 in healthy subjects. GSK2339345 is a blocker of neuronal voltage gated sodium channels in development for the treatment of chronic cough, excessive cough and post-viral and viral (acute) cough. Inhaled pan NaV inhibitors are associated with oropharyngeal sensation perturbation and so this study will establish the potential local sensate effects of GSK2339345 at multiples of the predicted inhaled therapeutic dose. This study also aims to define the maximum tolerated dose of GSK2339345.

Part A of this study will be conducted in healthy volunteers to investigate the safety and tolerability of GSK2339345, in particular examining oropharyngeal sensation perturbation. Part A is an open label, oral, single-dose escalating rinse, gargle and spit study. Assessments of sensate changes will include 4 point scale, assessment of sensation on base of tongue, sensation of temperature, assessment of taste, a water swallow test and assessment of potential paraesthesias. Part A will also include PK assessments to investigate the PK profile of GSK2339345.

Part B of this study is a randomised, double blind, placebo controlled, inhaled dose escalation study over two study days per dose to examine the possible adverse events such as transient mouth, throat and upper airway numbness in healthy volunteers. Similar assessments of sensations to those used in Part A will be performed. The potential for systemic cardiovascular (CV) or central nervous system (CNS) effects will also be assessed. Pharmacodynamic effects of GSK2339345 will be investigated in Part B using a capsaicin cough challenge. The study will investigate whether GSK2339345 can alter the capsaicin cough threshold (as determined by the capsaicin concentration required to induce 2 or more (C2) and 5 or more (C5) coughs) in healthy volunteers. Part B will also include PK assessments to investigate the PK profile of GSK2339345. Placebo will be used as a control and nebulised lidocaine will be used for control and blinding purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate Transaminase (AST), Alanine Transaminase (ALT), alkaline phosphatase and bilirubin ≤ 1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use an approved method of contraception, (double-barrier method or complete sexual inactivity by abstinence). This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Non-smoker for at least 6 months with a pack history ≤ 5pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight ≥ 50 kg and BMI within the range 19 - 32.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB< 450 msec
* A 24 hour Holter ECG at screening that demonstrates no clinically significant abnormalities or finding that could interfere with interpretation of the study results, when assessed by an appropriately trained and experienced reviewer.

Exclusion Criteria:

* Hepatitis B or Hepatitis C positive
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* HIV positive
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Forced Expiratory Volume in one second (FEV1) less than 80% of the predicted value prior to dosing (Part B only)
* Part B only: any subject who does not reach C5 following an oral inhalation challenge of capsaicin at a dose level of 250 μM at screening or Day -1, reaches C5 following an oral inhalation of placebo solution or has known hypersensitivity to capsaicin
* Part A only: any subject who is unable to gargle with placebo solution
* Any subject who is unable to perceive oropharyngeal numbness caused by lidocaine
* Any subject who, upon oropharyngeal examination, is deemed by the Investigator to be unsuitable for oropharyngeal sensation assessments. This includes any injuries to the mucosa of the mouth or pharynx that could potentially increase systemic absorption e.g candidiasis.
* Any patient with a history of swallowing difficulties.
* Any subject who has a history of an allergic reaction to a local anaesthetic. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Breath CO levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-17 (Actual); Primary Completion 2012-03-15 (Actual); Study Completion 2012-03-15 (Actual)

PRIMARY OUTCOMES:
Change in oropharyngeal sensation | Dosing to 1 hour post dose
  Measured by 4 point scale, fingertip electrode assessment, sensation to water temperature, adverse events, water swallow test and assessment of gag reflex
Adverse events (AEs) for all study participants | Dosing to 24 hours post dose
  Measurement of types of AEs reported, severity and relationship to study drug
Assessment of vital signs for all study participants | Screening to follow-up
  Triplicate measurements will be taken at screening and pre-dose, single measurements at all other timepoints
Holter ECG measurement for all study participants | Screening (Part A and Part B)
  24 hour Holter ECG will be taken at screening
12-lead ECG measurements for all study participants | Screening to follow-up
  Triplicate measurements will be taken at screening and pre-dose, single measurements at all other timepoints
Body temperature for all study participants | Screening, pre-dose, 30 mins post dose, 4 hours post dose, 8 hours post dose and follow-up in each dosing session
Safety laboratory assessments for all study participants | Part A: Screening, pre-dose, 24 hours post dose and follow-up in each dosing session. Part B: Screening, pre-dose and 8 hours post dose on Day 1, 0 hours and 8 hours post dose on Day 2, follow-up
  To include haematology and clinical biochemistry assessments
Cardiac troponin measurements for all study participants | Part B only: Screening, pre-dose and 24 hours post dose on Day 1

SECONDARY OUTCOMES:
Palatability by identification of solution taste and 11 point scale | 30 minutes post dose
Systemic pharmacokinetics of GSK2339345 using plasma concentrations of GSK2339345 and derived pharmacokinetic parameters | Pre-dose to 24 hours post dose
Effect of an inhaled nebulised dose of GSK2339345 on cough response to capsaicin challenge in healthy volunteers | Part B: Day 2, 10 minutes post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115419 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115419?search=study&search_terms=115419#rs
- Available data/document: Dataset Specification: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115419 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register